CLINICAL TRIAL: NCT05185856
Title: Visa-versa! Breaking Instead of Pushing the Pedals: Eccentric Exercise to Improve Training Performance in Patients With Chronic Lung Disease. A Single-center Randomized Controlled Trial
Brief Title: Visa-versa! Breaking Instead of Pushing the Pedals-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Visa-Versa!-B
Record Dates: First submitted 2021-12-06; First posted 2022-01-11 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Start with: Concentric (normal) cycling (Sham Comparator): Patients that are allocated to this arm will start with normal cycling
  Interventions: Procedure: 15 minutes eccentric cycling; Procedure: 15 minutes concentric (normal) cycling
- Start with: Eccentric cycling (Experimental): Patients that are allocated to this arm will start with eccentric cycling
  Interventions: Procedure: 15 minutes eccentric cycling; Procedure: 15 minutes concentric (normal) cycling

INTERVENTIONS:
Procedure: 15 minutes eccentric cycling — The exposure to eccentric exercise will be individualized-intensity stepwise incremental cycle exercise starting at 50 Watt with individually tailored increments every 5 minutes.
Procedure: 15 minutes concentric (normal) cycling — The exposure to concentric exercise will be individualized-intensity stepwise incremental cycle exercise starting at 50 Watt with individually tailored increments every 5 minutes.

SUMMARY:
Eccentric muscle work is defined as lengthening of a muscle while applying force. It was shown that with eccentric work, muscles are able to perform four times as much power compared to usual concentric work, which results in huge training gain with a highly decreased oxygen demand and thus lower cardiovascular load. Pulmonary hypertension (PH) is a chronic condition associated with significant reduced exercise capacity and increased morbidity and mortality, resulting in reduced quality of life. Physical training has been shown to be beneficial in PH, even in severely limited patients. However, due to cardiopulmonary constraints in PH, training intensities may be very low, so that many patients are physically almost unable to perform exercise on a high enough level to maintain muscle mass. A low body muscle not only feeds the vicious cycle of decreasing exercise capacity, but also has many deleterious metabolic and immunological consequences which further increase disability and decrease quality of life in PH. Thus, eccentric training, which allows to gain muscle mass with a low stress to the cardiopulmonary unit may to be highly beneficial for patients with PH and allied cardiopulmonary disease, such as chronic obstructive pulmonary disease (COPD) and heart failure. Therefore, the aim of the study is to compare differences in oxygen uptake (peak VO2 [l/min]) and other physiological measures during similar cardiopulmonary exercise test protocols of eccentric- vs. concentric cycling in PH- patients and comparators with or without other cardiopulmonary diseases.

DETAILED DESCRIPTION:
Eccentric muscle work is when a muscle lengthens while applying force. Although eccentric muscle work is part of everyday life, e.g. whilst descending, it is not integrated in modern training protocols and its underlying physiological mechanisms are still incompletely understood. It was shown that muscles are able to perform four times as much power eccentrically compared to common concentric muscle work with a comparably very low oxygen demand and thus cardiovascular load. Thus, eccentric training may be of special interest for patients with cardiopulmonary diseases. Since much higher training intensities are achieved eccentrically, the training increase after a few weeks of eccentric training is huge compared to ordinary concentric training. In addition, it has been observed that these high intensities applied eccentrically lead also to a concentric gain in strength and are therefore transferable to everyday activities. Physical training has been shown to be beneficial in almost every cardiovascular disease, even in severely limited patients. However, training intensities may be very low in some patients with advanced cardiopulmonary disease, so some patients are physically almost unable to perform exercise on a beneficial level. Thus, for this collective, eccentric training may to be a very intriguing option. Patients with pulmonary vascular diseases such as pulmonary arterial and chronic thromboembolic pulmonary hypertension (PH) per definition reveal an elevated pulmonary artery pressure (PAP) along with an increased pulmonary vascular resistance (PVR). However, also other common diseases, such as left heart disease (LHD) or chronic obstructive pulmonary disease (COPD) are often associated with PH. The cardinal symptoms of PH is dyspnea on exertion leading to limited exercise performance, daily activity and quality of life. PH-patients also benefit from structured exercise training, but training intensities might be limited in patients with advanced disease. A few studies have investigated eccentric exercising in cardiopulmonary patients but none in PH. Most of these studies are in patients with coronary heart disease- (CHD) or COPD, including only few participants and often studies did not followed sound methodologies, such as randomized-controlled trial (RCT) protocols However, even in the hitherto limited patients´ investigated, eccentric training was assessed beneficial, feasible and safe.

The physiological cardiopulmonary response to eccentric exercising has not been investigated in patients with PH and the physiological basis to investigate such training opportunities is completely lacking.

The aim of this project is to investigate the cardiopulmonary effects of eccentric exercise in using solid randomized-controlled research protocols in cardiopulmonary diseases with focus on PH in order to provide a basis to the question of whether this promising training method could become established in cardiopulmonary rehabilitation, especially in patients with advanced disease and pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* In a stable condition on the same disease specific medication >4 weeks.
* Signed informed consent.
* Patients with chronic obstructive pulmonary (COPD) with a FEV1/FVC-ratio > 0.7

Exclusion Criteria:

* Severe daytime hypoxemia (pO2 ≤7.3 kPa or <55 mmHg).
* Other clinically significant concomitant disease states (e.g., renal, hepatic dysfunction, etc.).
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorder, dementia or confusional state of the subject, neurological or orthopedic problems with inability to ride a bicycle.
* Woman with known pregnancy (Women with known pregnancy will not be allowed into the study. It will however not be searched for early unknown pregnancy in woman of child-bearing potential, as cycling is not contraindicated in early unknown pregnancy stage and we thus do not plan routine pregnancy tests before study entrance in women of childbearing potential).
* Enrolment into another clinical trial with active treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Oxygen uptake (peak VO2 [l/min]) | 1 Day
  Difference in oxygen uptake (peak VO2 [l/min]) of eccentric vs. concentric cycling exercise.

SECONDARY OUTCOMES:
Respiratory exchange ratio (RER) | 1 day
  Volume carbon dioxide devided by the volume of oxygen( VCO2/VO2)
Breathing equivalent for carbon dioxide | 1 day
  Minute ventilation divided by volume carbon dioxide (VE/VCO2)
Pulmonary end tidal carbon dioxide (PET CO2) | 1 day
  The level of carbon dioxide that is released at the end of an exhaled breath
Arterial oxygen saturation (SpO2) | 1 day
  Noninvasively measured oxygenation of the hemoglobin by pulse oximetry (Light Sensors)
Borg Scale for dyspnea | 1 day
  Patient reported level of dyspnea on the Borg Scale from minimum 0 to maximum 10 while 10 is the worst dyspnea and 0 is no dyspnea.
Borg Scale for leg fatigue | 1 day
  Patient reported level of leg fatigue on the Borg Scale from minimum 0 to maximum 10 while 10 is the worst leg fatigue and 0 i no leg fatigue.
Cardiac output | 1 day
  How many liters blood is the heart able to move in one minute. Assessed by echocardiography.
Pulmonary Artery Pressure | 1 day
  Right ventricle pressure divided by the right atrium pressure gradient (RV/RA pressure gradient) to assess the systolic pulmonary artery pressure by echocardiography
Blood pressure | 1 day
  Systolic and diastolic blood pressure assessed by arm cuff measurement
Brain tissue oxygenation | 1 day
  Oxygenation of the brain tissue assessed by light sensors on the forehead
Muscle tissue oxygenation | 1 day
  Oxygenation of the muscle tissue assessed by light sensors on the quadriceps muscle
Arterial blood gases: PH | 1 day
  Arterial blood gases: PH, assessed by arterial blood sample
Arterial blood gases: Partialpressure for oxygen (PaO2) | 1 day
  Arterial blood gases: Partialpressure for oxygen (PaO2), assessed by arterial blood sample
Arterial blood gases: Bicarbonate (HCO3) | 1 day
  Arterial blood gases: Bicarbonate (HCO3), assessed by arterial blood sample
Arterial blood gases: lactate | 1 day
  Arterial blood gases: lactate, assessed by arterial blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No